CLINICAL TRIAL: NCT00723398
Title: Combination of Low Dose Antiestrogens With Omega-3 Fatty Acids for Prevention of Hormone-independent Breast Cancer
Brief Title: Nutritional Supplements and Hormonal Manipulations for Breast Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Andrea Manni, Professor and Chief Division of Endocrinology, Diabetes, and Metabolism, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 26970
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Breast Cancer
Keywords: omega-3 fatty acids; antiestrogens; breast cancer prevention; breast density; biomarkers of mammary carcinogenesis
MeSH Terms: conditions — Breast Neoplasms | interventions — Raloxifene Hydrochloride; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Group 1: Control (No Intervention): Control, no intervention
- Group 2: Raloxifene 60 Mg Oral Tablet (Experimental): Raloxifene 60 mg Orally Daily
  Interventions: Drug: Raloxifene 60 Mg Oral Tablet
- Group 3: Raloxifene 30 Mg Oral Tablet (Experimental): Raloxifene 30 mg Orally Daily
  Interventions: Drug: Raloxifene 30 Mg Oral Tablet
- Group 4: Lovaza 4 gm oral (Experimental): Lovaza 4 gm/day Orally with Meals
  Interventions: Dietary Supplement: Lovaza 4gm oral
- Group 5: Lovaza 4gm & Raloxifene 30mg (Experimental): Lovaza 4 gm/day oral capsule with meals plus Raloxifene 30 mg oral tablet daily
  Interventions: Drug: Lovaza 4gm & Raloxifene 30mg

INTERVENTIONS:
Dietary Supplement: Lovaza 4gm oral — Dietary supplement; Take 4 mg oral capsules daily
  Other Names: Omega-3 Fatty Acid Capsules; Fish Oil capsules; Triklo
  Arms: Group 4: Lovaza 4 gm oral
Drug: Raloxifene 60 Mg Oral Tablet — 60 mg orally every day for two years
  Other Names: Evista 60 Mg Oral Tablet
  Arms: Group 2: Raloxifene 60 Mg Oral Tablet
Drug: Raloxifene 30 Mg Oral Tablet — 30 mg orally daily for two years
  Other Names: Evista 30 Mg Oral Tablet
  Arms: Group 3: Raloxifene 30 Mg Oral Tablet
Drug: Lovaza 4gm & Raloxifene 30mg — Lovaza 4gm and Raloxifene 30 Mg orally once per day for 2 years
  Other Names: Pitavastatin 4 gm and Evista 30 mg oral tablet
  Arms: Group 5: Lovaza 4gm & Raloxifene 30mg

SUMMARY:
The overall hypothesis is that the combination of a low dose of the antiestrogen Raloxifene with omega-3 fatty acids will exert a synergistic breast cancer chemopreventive effect due to the crosstalk of their downstream cellular effects leading to decreased proliferation and increased apoptosis of premalignant mammary cells. Based on the investigators hypothesis that upregulation of functional estrogen receptors in the premalignant lesions is also responsible for the development of hormone independent tumors, the investigators postulate that the combination of antiestrogens and omega-3 fatty acids will reduce the development of both hormone-dependent and -independent tumors. At present, there are no known interventions able to decrease the development of hormone-independent tumors, which are more prevalent, more aggressive, leading to the patient's demise. In addition, the investigators postulate that this approach will be safe since it will combine a lower and hence a less toxic dose of Raloxifene with the administration of omega-3 fatty acids which are known to have health benefits, i.e., reduction in cardiovascular risk, beyond their possible chemo preventive effect in breast cancer.

DETAILED DESCRIPTION:
The main objectives of this study are to determine the individual and combined effects of Raloxifene and omega-3 fatty acids on surrogate markers of breast cancer development in healthy, postmenopausal women. The primary endpoint will be mammographic density for which the study has been powered. Breast density is a major risk factor for breast cancer and hence it is chosen to evaluate the potential chemopreventive efficacy of our interventions. Secondary endpoints would include markers of oxidative stress, parameters of estrogen metabolism, markers of inflammation, and markers of IGF-I signaling, all of which have been shown in the literature to have an influence on mammary carcinogenesis.

Study Population: Healthy, postmenopausal women between the ages of 35-70 years, undergoing yearly mammograms as part of routine screening practice.

Method of Identification of Subjects/Samples/Medical Records: Women reporting for yearly mammograms will be considered for this protocol. They will be given first a screening questionnaire to rule out any co-existing medical condition that would predispose them to thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status defined as history of at least 12 months without spontaneous menstrual bleeding or a documented hysterectomy and bilateral salpingo oophorectomy
* Breast density greater than 25%
* No hormone replacement therapy for at least six months prior to entry into this study
* Non-smokers.

Exclusion Criteria:

* History of stroke, pulmonary embolism or deep vein thrombosis
* History of atherosclerotic heart disease
* Presence of any known hypercoagulable state either congenital (e.g., protein S deficiency) or acquired (e.g., corticosteroid treatment)
* Diabetes mellitus
* Uncontrolled hypertension (BP ≥140/90)
* Presence of a psychiatric condition that would interfere with adherence to the protocol.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Manni, MD, Principal Investigator — Penn State University
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manni A, Richie JP, Schetter SE, Calcagnotto A, Trushin N, Aliaga C, El-Bayoumy K. Stearoyl-CoA desaturase-1, a novel target of omega-3 fatty acids for reducing breast cancer risk in obese postmenopausal women. Eur J Clin Nutr. 2017 Jun;71(6):762-765. doi: 10.1038/ejcn.2016.273. Epub 2017 Feb 1. PMID 28145413

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: Raloxifene 60 mg: Raloxifene 60 mg Orally Daily
- Group 3: Raloxifene 30 mg: Raloxifene 30 mg Orally Daily
- Group 4: Lovaza 4 gm: Lovaza 4 gm/day Orally with Meals
- Group 5: Lovaza 4 gm and Raloxifene 30 mg: Lovaza 4 gm/day orally with meals plus Raloxifene 30 mg orally daily
Period: Overall Study
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Started | 53 | 53 | 53 | 54 | 53
Completed | 47 | 38 | 36 | 49 | 44
Not Completed | 6 | 15 | 17 | 5 | 9
Not completed — Withdrawal by Subject | 2 | 6 | 4 | 4 | 4
Not completed — Protocol Violation | 2 | 1 | 5 | 0 | 0
Not completed — Physician Decision | 2 | 2 | 5 | 0 | 1
Not completed — Adverse Event | 0 | 5 | 3 | 1 | 4
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg | Total
Number analyzed (Participants) | 53 | 53 | 53 | 54 | 53 | 266
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 49 | 43 | 48 | 45 | 46 | 231
  >=65 years | 4 | 10 | 5 | 9 | 7 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 53 | 53 | 54 | 53 | 266
  Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 52 | 53 | 53 | 53 | 53 | 264
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 1 | 1 | 1 | 0 | 4
  White | 51 | 52 | 52 | 51 | 53 | 259
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute Breast Density
Description: Change of absolute breast density as indicated by mammography from baseline to Year +1 and completion of study (Year +2). No other mammograms will be obtained or used for the purpose of this study. Absolute breast density volume is based on breast thickness and the x-ray attenuation at each pixel of the image.
Time Frame: 2 years
Population: The decrease in the population groups is accounted for through subject withdrawals, subjects lost to follow-up, and other reasons for not completing study.
Measure: Mean (Standard Deviation); unit: cm squared
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 53 | 53 | 53 | 54 | 53
cm squared
  Absolute density at baseline | 65.53 (59.43) | 64.39 (39.95) | 65.08 (34.47) | 56.35 (22.61) | 63.81 (29.81)
  Absolute density at 1 year: number analyzed (Participants) | 48 | 41 | 41 | 50 | 45
  Absolute density at 1 year | 59.29 (40.72) | 60.48 (38.89) | 59.53 (30.32) | 58.87 (22.21) | 60.93 (24.64)
  Absolute density at 2 years: number analyzed (Participants) | 46 | 38 | 37 | 48 | 44
  Absolute density at 2 years | 54.34 (20.11) | 60.57 (35.10) | 58.86 (27.93) | 57.60 (20.77) | 28.53 (25.18)

2. Secondary Outcome: Changes in Biomarkers for Oxidative Stress:Urinary 8-(Isoprostane) F-2α
Description: Changes in biomarkers for oxidative stress. Specific time points for evaluation are baseline and Year +1 (only). Urinary 8-(isoprostane) F-2α as measured through urine analysis.
Time Frame: 1 year
Population: Biomarker measurements were not taken for the entire population of the study due to non-significant trends for treatment effects found in this population (n = 47).
Measure: Mean (Standard Error); unit: pg/mg creatinine
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 8 | 10 | 10 | 11 | 8
pg/mg creatinine
  Baseline | 544 (105) | 366 (39.7) | 530 (107) | 440 (30.8) | 444 (54.6)
  1 year | 484 (77.3) | 360 (33.8) | 538 (67.0) | 313 (45.1) | 396 (40.6)

3. Secondary Outcome: Changes in Biomarkers for Oxidative Stress: Urinary 8-hydroxy-deoxyguansine
Description: Changes in biomarkers for oxidative stress. Specific time points for evaluation are baseline and Year +1 (only). Urinary 8-hydroxy-deoxyguansine as measured through urinary analysis.
Time Frame: 1 year
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mg creatinine
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 8 | 10 | 10 | 11 | 8
ng/mg creatinine
  Baseline | 255 (63.6) | 285 (47.7) | 213 (91.0) | 184 (25.6) | 355 (79.7)
  1 year | 224 (31.8) | 309 (69.0) | 246 (108) | 177 (17.3) | 297 (90.2)

4. Secondary Outcome: Changes in Biomarkers for Estrogen Metabolism: 2-hydroxy Estrone (Urinary 2-OHE1) and 16-α-hydroxy Estrone (16α-OHE1)
Description: Changes in biomarkers for estrogen metabolism: 2-hydroxy estrone (Urinary 2-OHE1) and 16-α-hydroxy estrone (16α-OHE1) as measured by urinary analysis. Specific time points for evaluation are baseline and Year +1 (only).
Time Frame: 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mg creatinine
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 8 | 10 | 10 | 11 | 8
ng/mg creatinine
  Baseline: Urinary 2-OHE1 | 10.57 (2.3) | 8.58 (1.0) | 8.82 (1.4) | 7.15 (1.1) | 15.6 (4.5)
  1 year: Urinary 2-OHE1 | 7.46 (1.4) | 10.03 (1.0) | 9.10 (1.4) | 7.49 (1.0) | 13.2 (3.7)
  Baseline: 16α-OHE1 | 6.22 (0.7) | 5.08 (0.5) | 6.86 (1.8) | 5.24 (0.5) | 6.6 (0.9)
  1 year: 16α-OHE1 | 5.68 (0.7) | 4.35 (0.5) | 7.46 (1.4) | 4.79 (0.3) | 5.68 (0.9)

5. Secondary Outcome: Changes in Serum Biomarkers for Inflammation From Levels of High Sensitivity C-reactive Protein (hsCRP) and Interleukin 6 (IL-6)
Description: Changes in serum biomarkers for inflammation including highly sensitive C-reactive protein and IL-6 obtained through a blood draw. Specific time points for evaluation are baseline and Year +1 (only).
Time Frame: 1 Year
Population: Biomarker measurements were not taken for the entire population of the study (N = 266) due to non-significant trends for treatment effects found in this initial population (n = 89).
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 17 | 17 | 18 | 21 | 16
pg/ml
  Baseline: Serum hsCRP | 2.39 (0.87) | 0.91 (0.26) | 1.67 (0.63) | 1.22 (0.31) | 4.28 (1.61)
  1 year: Serum hsCRP | 2.19 (0.63) | 1.04 (0.34) | 1.34 (0.34) | 1.69 (0.59) | 2.59 (0.89)
  Baseline: Serum IL-6: number analyzed (Participants) | 8 | 10 | 10 | 11 | 8
  Baseline: Serum IL-6 | 1.27 (0.3) | 1.14 (0.23) | 1.04 (0.22) | 1.32 (0.45) | 1.84 (0.52)
  1 year: Serum IL-6: number analyzed (Participants) | 8 | 10 | 10 | 11 | 8
  1 year: Serum IL-6 | 1.03 (0.19) | 1.13 (0.26) | 1.11 (0.2) | 1.49 (0.41) | 1.32 (0.34)

6. Secondary Outcome: Changes in Insulin-like Growth Factor-1 (IGF-1) and Insulin-like Growth Factor-1 Binding Protein-3 (IGFBP-3)
Description: Changes in insulin-like growth factor-1 (IGF-1) and insulin-like growth factor-1 binding protein-3 (IGFBP-3) obtained through blood sample. Specific time points for evaluation are baseline and Year +1 (only).
Time Frame: 1 year
Population: Measurements were not taken for the entire population of the study due to non-significant trends for treatment effects found in this population (n = 46).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 8 | 9 | 10 | 11 | 8
ng/mL
  Baseline: IGF-1 | 4.96 (0.37) | 4.63 (0.28) | 4.80 (0.23) | 4.95 (0.41) | 4.89 (0.49)
  1 year: IGF-1 | 5.05 (0.44) | 4.40 (0.25) | 4.76 (0.24) | 4.96 (031) | 4.82 (0.52)
  Baseline: IGFBP-3 | 7.67 (0.32) | 7.53 (0.19) | 7.69 (0.21) | 7.83 (0.20) | 7.57 (0.23)
  1 year: IGFBP-3 | 7.75 (0.26) | 7.55 (0.12) | 7.79 (0.24) | 7.83 (0.17) | 7.61 (0.23)

7. Secondary Outcome: Changes in Serum Lipid Levels
Description: Changes in serum lipid levels as measured through total cholesterol, low-density lipoprotein (LDL) cholesterol, high-density lipoprotein (HDL) cholesterol, and triglycerides. Specific time points for evaluation are baseline, Year +1, and Year 2.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 53 | 51 | 52 | 54 | 52
mg/dL
  Baseline: Total Cholesterol | 207.3 (41.18) | 203.6 (29.98) | 204.3 (36.29) | 197.7 (33.2) | 197.6 (38.68)
  1 year: Total Cholestrol: number analyzed (Participants) | 48 | 42 | 41 | 51 | 45
  1 year: Total Cholestrol | 208.8 (34.39) | 198.3 (29.33) | 199.6 (28.43) | 199.6 (30.45) | 189.4 (33.45)
  2 year: Total Cholesterol: number analyzed (Participants) | 47 | 38 | 36 | 49 | 44
  2 year: Total Cholesterol | 207.5 (36.41) | 196.6 (30.64) | 202.3 (25.58) | 200.2 (34.55) | 192.6 (30.02)
  Baseline: LDL Cholesterol | 114 (38.07) | 114.7 (27.53) | 111.2 (31.83) | 106.6 (31.96) | 108.1 (35.87)
  1 year: LDL Cholesterol: number analyzed (Participants) | 48 | 42 | 41 | 51 | 45
  1 year: LDL Cholesterol | 115.1 (31.99) | 106.8 (25.98) | 106.2 (24.38) | 109.7 (29.22) | 96.58 (26.37)
  2 year: LDL Cholesterol: number analyzed (Participants) | 47 | 38 | 36 | 49 | 44
  2 year: LDL Cholesterol | 115.3 (29.21) | 104.7 (28.13) | 106.1 (25.4) | 110.4 (29.2) | 99.48 (25.2)
  Baseline: HDL Cholesterol | 68.75 (18.83) | 66.18 (15.47) | 70.92 (18.54) | 68.06 (16.89) | 68.9 (17.68)
  1 year: HDL Cholesterol: number analyzed (Participants) | 48 | 42 | 41 | 51 | 45
  1 year: HDL Cholesterol | 70.71 (18.87) | 68.88 (14.06) | 70.59 (16.63) | 70.59 (18.31) | 76.11 (18.61)
  2 year: HDL Cholestrol: number analyzed (Participants) | 47 | 38 | 36 | 49 | 44
  2 year: HDL Cholestrol | 70.19 (19.35) | 68.63 (15.04) | 73.17 (18.01) | 70.67 (19.38) | 75.77 (17.8)
  Baseline: Triglycerides | 122.7 (54.57) | 113.2 (48.39) | 110.6 (50.49) | 115.1 (52.33) | 103.6 (38.79)
  1 year: Triglycerides: number analyzed (Participants) | 48 | 42 | 41 | 51 | 45
  1 year: Triglycerides | 114.5 (62.95) | 113.2 (55.08) | 113.7 (49.76) | 96.22 (42.94) | 83.71 (31.08)
  2 year: Triglycerides: number analyzed (Participants) | 47 | 38 | 36 | 49 | 44
  2 year: Triglycerides | 110.1 (44.25) | 116.9 (50.17) | 115.8 (58.48) | 95.41 (49.6) | 86.43 (35)

8. Secondary Outcome: Changes in Complete Blood Count: Red Blood Cells
Description: Changes in complete blood count levels as measured through red blood cells (RBC). Specific time points for evaluation are baseline, Year +1, and Year 2.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millions of cells per microliter
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 53 | 51 | 50 | 51 | 50
millions of cells per microliter
  Baseline: RBC | 4.31 (0.33) | 4.25 (0.30) | 4.30 (0.33) | 4.33 (0.43) | 4.24 (0.31)
  1 year: RBC: number analyzed (Participants) | 48 | 42 | 41 | 50 | 45
  1 year: RBC | 4.27 (0.32) | 4.19 (0.25) | 4.25 (0.30) | 4.36 (0.44) | 4.20 (0.32)
  2 year: RBC: number analyzed (Participants) | 46 | 38 | 35 | 49 | 44
  2 year: RBC | 4.32 (0.36) | 4.20 (0.23) | 4.24 (0.35) | 4.33 (0.45) | 4.23 (0.31)

9. Secondary Outcome: Changes in Complete Blood Count: Hemoglobin
Description: Changes in complete blood count levels as measured through hemoglobin. Specific time points for evaluation are baseline, Year +1, and Year 2.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 53 | 51 | 50 | 51 | 50
g/dL
  Baseline: Hemoglobin | 13.09 (1.56) | 13.11 (1.48) | 12.73 (2.02) | 13.25 (0.99) | 13.35 (0.86)
  1 year: Hemoglobin: number analyzed (Participants) | 48 | 42 | 41 | 50 | 45
  1 year: Hemoglobin | 12.97 (1.49) | 12.97 (1.61) | 12.95 (0.96) | 13.33 (0.97) | 13.10 (1.65)
  2 year: Hemoglobin: number analyzed (Participants) | 46 | 38 | 35 | 49 | 44
  2 year: Hemoglobin | 13.10 (0.87) | 13.07 (0.71) | 12.82 (0.96) | 13.16 (0.91) | 13.22 (0.95)

10. Secondary Outcome: Changes in Complete Blood Count: Hematocrit
Description: Changes in complete blood count levels as measured through hematocrit percentage. Specific time points for evaluation are baseline, Year +1, and Year 2.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: volume percentage
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 53 | 51 | 50 | 51 | 50
volume percentage
  Baseline: Hematocrit | 39.14 (2.50) | 38.95 (2.49) | 38.79 (3.06) | 39.09 (2.70) | 39.20 (2.48)
  1 year: Hematocrit: number analyzed (Participants) | 48 | 42 | 41 | 50 | 45
  1 year: Hematocrit | 38.83 (2.25) | 38.79 (2.14) | 38.43 (2.69) | 39.52 (2.72) | 39.14 (2.52)
  2 year: Hematocrit: number analyzed (Participants) | 46 | 38 | 35 | 49 | 44
  2 year: Hematocrit | 39.00 (2.47) | 38.86 (2.28) | 38.31 (2.84) | 38.59 (5.72) | 39.14 (2.74)

11. Secondary Outcome: Changes in Complete Blood Count: White Blood Cells and Platelets
Description: Changes in complete blood count levels as measured through white blood cells (WBC) and platelets. Specific time points for evaluation are baseline, Year +1, and Year 2.
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: thousand cells/mL
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Number analyzed (Participants) | 53 | 51 | 50 | 51 | 50
thousand cells/mL
  Baseline: WBC: number analyzed (Participants) | 52 | 51 | 50 | 51 | 50
  Baseline: WBC | 5.13 (1.29) | 5.47 (1.57) | 5.00 (1.20) | 5.04 (1.64) | 5.27 (1.24)
  1 year: WBC: number analyzed (Participants) | 48 | 42 | 41 | 50 | 45
  1 year: WBC | 5.15 (1.76) | 5.51 (1.54) | 4.78 (1.04) | 4.95 (1.37) | 4.91 (1.18)
  2 year: WBC: number analyzed (Participants) | 46 | 38 | 35 | 49 | 44
  2 year: WBC | 5.14 (1.32) | 5.42 (1.39) | 4.90 (1.10) | 4.90 (1.26) | 4.91 (1.19)
  Baseline: Platelets: number analyzed (Participants) | 53 | 50 | 50 | 51 | 50
  Baseline: Platelets | 270.70 (277.46) | 235.22 (52.06) | 240.42 (41.32) | 237.33 (51.41) | 235.76 (53.07)
  1 year: Platelets: number analyzed (Participants) | 48 | 42 | 41 | 50 | 45
  1 year: Platelets | 237.02 (55.05) | 228.02 (50.71) | 230.61 (39.40) | 231.42 (49.58) | 221.49 (55.50)
  2 year: Platelets: number analyzed (Participants) | 46 | 38 | 35 | 49 | 44
  2 year: Platelets | 234.02 (47.55) | 226.16 (51.14) | 232.09 (44.10) | 232.47 (54.22) | 223.27 (49.18)

ADVERSE EVENTS:
Time Frame: Participants who did not meet an off study criterion were followed until 2 years post initiation of the study medication regimen.
Arm/Group | Group 1: Control | Group 2: Raloxifene 60 mg | Group 3: Raloxifene 30 mg | Group 4: Lovaza 4 gm | Group 5: Lovaza 4 gm and Raloxifene 30 mg
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/53 | 0/53 | 0/54 | 0/53
Other Adverse Events (participants affected / at risk) | 1/53 | 10/53 | 7/53 | 0/54 | 6/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Control (N=53) | Group 2: Raloxifene 60 mg (N=53) | Group 3: Raloxifene 30 mg (N=53) | Group 4: Lovaza 4 gm (N=54) | Group 5: Lovaza 4 gm and Raloxifene 30 mg (N=53)
Endometrial Cancer (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Endometrial Cancer (unlikely a secondary malignancy- likely new primary)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Control (N=53) | Group 2: Raloxifene 60 mg (N=53) | Group 3: Raloxifene 30 mg (N=53) | Group 4: Lovaza 4 gm (N=54) | Group 5: Lovaza 4 gm and Raloxifene 30 mg (N=53)
Hot flashes (Endocrine disorders) | 0 (0) | 10 (10) | 7 (7) | 0 (0) | 6 (6)
Night Sweating (diaphoresis) (General disorders) | 0 (0) | 6 (6) | 3 (3) | 0 (0) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Vaginal Spotting (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Leg cramping (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes